CLINICAL TRIAL: NCT00485394
Title: A Randomized, Double-Masked, Dose-Ranging, Multi-Center, Phase II Study Comparing the Safety and Efficacy of OT-551 With Placebo to Treat Geographic Atrophy Associated With Age-Related Macular Degeneration
Brief Title: The OMEGA Study: Use of Eye Drops to Treat Geographic Atrophy Associated With Age-Related Macular Degeneration (Dry AMD)
Acronym: OMEGA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Othera Pharmaceuticals (Industry)
Responsible Party: Alison Brown, Othera Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OT-551-C04
Record Dates: First submitted 2007-06-11; First posted 2007-06-13 (Estimated); Last update posted 2008-04-02 (Estimated); Status verified 2008-03

CONDITIONS: Age-Related Macular Degeneration
Keywords: AMD; age-related macular degeneration; geographic atrophy; GA
MeSH Terms: conditions — Macular Degeneration; Geographic Atrophy | interventions — OT-551

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): OT-551 0.3% ophthalmic solution
  Interventions: Drug: OT-551
- 2 (Experimental): OT-551 0.45% ophthalmic solution
  Interventions: Drug: OT-551
- 3 (Placebo Comparator): vehicle placebo
  Interventions: Drug: vehicle placebo

INTERVENTIONS:
Drug: OT-551 — OT-551 0.3% ophthalmic solution, 2 drops 4 times daily
  Arms: 1
Drug: OT-551 — OT-551 0.45% ophthalmic solution, 2 drops 4 times daily
  Arms: 2
Drug: vehicle placebo — OT-551 0% ophthalmic solution, 2 drops 4 times daily
  Arms: 3

SUMMARY:
The purpose of this trial is to compare the ability of two doses of OT-551 ophthalmic solution and drug-free solution to safely and effectively treat geographic atrophy associated with age-related macular degeneration.

DETAILED DESCRIPTION:
Age-related macular degeneration (AMD) results in severe, irreversible central vision loss and is the leading cause of blindness in individuals older than 50 years in the western world. The vast majority of AMD patients have the 'dry' (non-exudative) form that is characterized by the presence of drusen and atrophic changes in the retinal pigment epithelium (RPE). Dry AMD may remain static or progress slowly to produce areas of geographic atrophy (GA), the advanced or late-stage form of dry AMD. GA is a severe vision-threatening lesion of the macula that may impair visual function, impact daily life activities, and result in blindness. Currently, there is no approved treatment for dry AMD or GA. Pre-clinical results have shown that OT-551 may protect RPE cells and photoreceptors from oxidative damage and block angiogenesis stimulated by VEGF and other growth factors, and therefore is a therapeutic candidate for treating GA.

ELIGIBILITY:
Inclusion Criteria:

* have a clinical diagnosis of GA in one or both eyes;
* be of non-childbearing potential

Exclusion Criteria:

* have GA secondary to any condition other than AMD in the study eye;
* have a BCVA of 20/200 or worse in the non-study eye;
* have a history of or current choroidal neovascularization in either eye, or the need for any study eye anti-angiogenic therapy;
* have any ocular condition in the study eye that would progress during the course of the study and could affect central vision or other ocular conditions that may be a confounding factor in this study;
* need to wear contact lenses in the study eye during the study;
* had confounding ocular surgery in the study eye;
* have concomitant treatment with any systemic or ocular medication that is known to be toxic to the lens, retina, or optic nerve;

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2007-06; Primary Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
Change in the area of GA | 2 years

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Mesa, Arizona
  - Tucson, Arizona
  - Beverly Hills, California
  - Oxnard, California
  - Sacramento, California
  - Denver, Colorado
  - Boynton Beach, Florida
  - Miami, Florida
  - Indianapolis, Indiana
  - Novi, Michigan
  - New York, New York
  - Charlotte, North Carolina
  - Cleveland, Ohio
  - Lakewood, Ohio
  - Portland, Oregon
  - Dallas, Texas
  - Houston, Texas

REFERENCES:
- See also: Othera Pharmaceuticals, Inc. website — http://www.othera.com